CLINICAL TRIAL: NCT04239066
Title: Penile Ischemia for Hypospadias Repair and The Patients and Surgeons Reported Outcomes. A Prospective Randomized Study
Brief Title: Penile Ischemia for Hypospadias Repair and The Patients and Surgeons Reported Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOURNIQUE.HYPOSPADIAS
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hypospadias; Hypospadias, Coronal; Hypospadia, Repair; Tourniquet
Keywords: Tourniquet; Hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Tourniquets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tourniquet (Experimental): tubularized incided plate (TIP) urethroplasty plus tourniquet
  Interventions: Procedure: Tourniquet
- Non-tourniquet (Experimental): tubularized incided plate (TIP) urethroplasty plus non-tourniquet
  Interventions: Procedure: Non-tourniquet

INTERVENTIONS:
Procedure: Tourniquet — tubularized incided plate (TIP) urethroplasty plus tourniquet
  Arms: Tourniquet
Procedure: Non-tourniquet — tubularized incided plate (TIP) urethroplasty plus non-tourniquet
  Arms: Non-tourniquet

SUMMARY:
Although haemostasis aimed to maintain bloodless surgical field for better exposure for the surgeon, cosmetic impact, and decreased breakdown of repair, there is no trials regarding the impact of haemostasis techniques on surgeon satisfaction during surgery and patients reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* distal penile hypospadias were eligible for tubularized incided plate (TIP) urethroplasty repair

Exclusion Criteria:

* coagulopathy
* sickle cell disease or sickle cell trait
* circumcised patient
* history of previous failed surgery
* severe chordee (>30 degree after degloving).

Ages: 6 Months to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
assess Intraoperative blood loss | 12 months
  by blood loss in milliliter in used gauze piece
bipolar diathermy use | 12 months
  by number of bipolar diathermy usage
Surgeon satisfaction about haemostasis | 12 months
  Surgeon satisfaction 4-tiered questionnaire (very satisfied, satisfied, unsatisfied and very unsatisfied).

SECONDARY OUTCOMES:
Patient-reported satisfaction | 24 months
  by hypospadias objective scoring evaluation (HOSE) questionnaire
Long term complication rate | 60 months
  number of surgery related complication after 5 years post operative

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Dawaba, PhD, Study Director — Mansoura University
Locations (1):
- Urology and nephrology center, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: Undecided